CLINICAL TRIAL: NCT04534166
Title: A Model for Risk Prediction of Fracture in Diabetic Patients With Osteoporosis
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-20-020
Record Dates: First submitted 2020-08-26; First posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Healthcare; Risk Prediction; Diabetic Patients With Osteoporosis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Risk Prediction of Fracture in Diabetic Patients with Osteoporosis — Risk Prediction of Fracture in Diabetic Patients with Osteoporosis

SUMMARY:
The fracture risk of diabetic patients proves to be higher than those without diabetesdue to thehyperglycemia, usage of diabetes drugs, the changes in insulin levels and excretion, and this risk begins as early as adolescence.Many factors may be related to bone metabolism in patients with diabetes, including demographic data (e.g. age, height, weight, gender), medical history (e.g. smoking, drinking, menopause) and examination (e.g. bone mineral density, blood routine), urine routine).However, most of existing methods are qualitative assessments and do not take the interactions of the physiological factors of humans into consideration. In addition, the fracture risk of diabetic patients with osteoporosis has not been further studied before. In order to investigate the effect of patients' physiological factors on fracture risk, in the paper, we used a hybrid model combining XGBoost with deep neural network to predict the fracture risk of diabetic patients with osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients in Hospital's outpatient and inpatient His database between July 2012 and November 2022, diabetic patients were combined with osteoporosis.

Exclusion Criteria:

* Patients with fractures before diagnosis of diabetes; patients with fractures before diagnosis of osteoporosis; patients with hyroid disease and other diseases that seriously affect bone metabolism.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chinese
Sampling Method: Non-Probability Sample
Dates: Start 2012-07-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Fracture | 2-10 year

IPD SHARING:
Plan to Share IPD: Undecided